CLINICAL TRIAL: NCT03776916
Title: Optimization of Simethicone Administration Strategy Before Esophagogastroscopy
Brief Title: Application of Simethicone in Esophagogastroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 307-simethicone
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-05

CONDITIONS: Gastric Disease
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Simethicone administration 20-30 min before the procedure:
  Patients intake simethicone solution 20-30 min before the procedure.
  Interventions: Other: Simethicone administration 20-30 min before the procedure
- Group 2 (Experimental): Simethicone administration 31-60 min before the procedure:
  Patients intake simethicone solution 31-60 min before the procedure.
  Interventions: Other: Simethicone administration 31-60 min before the procedure
- Group 3 (Experimental): Simethicone administration >60 min before the procedure; Patients intake simethicone solution >60 min before the procedure.
  Interventions: Other: Simethicone administration > 60 min before the procedure

INTERVENTIONS:
Other: Simethicone administration 20-30 min before the procedure — Patients intake simethicone 20-30 min before the procedure
  Arms: Group 1
Other: Simethicone administration 31-60 min before the procedure — Patients intake simethicone administration 31-60 min before the procedure.
  Arms: Group 2
Other: Simethicone administration > 60 min before the procedure — Patients intake simethicone administration > 60 min before the procedure.
  Arms: Group 3

SUMMARY:
This is a randomized controlled trial to comparing the different simethicone administration strategies for esophagogastroscopy. Recent studies have indicated that the administration of simethicone before endoscopic examination could shorten the procedure time and improve the diagnostic rate of the gastric mucosal lesions. But the time interval between simethicone administration and the examination has not been fully determined. This study will test whether the time of taking simethicone before endoscopy could influence the performance of the procedure in a randomized controlled trial. The results may benefit the current clinical practice.

DETAILED DESCRIPTION:
Esophagogastroscopy can enable the direct examination of the esophageal and gastric mucosal lesions, which has been widely applied in clinical practice. However, during the examination, too much water, foam or residues in the stomach will not only increase the procedure time and the misdiagnosis rate, but also decrease the patients' tolerance, for more efforts should be made to deal with the excessive water, foam or residues in order to obtain a clear view of the mucosa. Simethicone is also called poly-dimethylsiloxane, which can be used to remove the foam and water. Although simethicone has been routinely administrated before the esophagogastroscopy, the optimal strategy of administrating simethicone has not been clearly investigated, especially the time to administrate simethicone. Intaking simethicone too early will result in too excessive water in the stomach, while if the patients take it too late it doesn't take effects. Thus, this is a study to determine whether selecting different simethicone administration strategies could improve the performance of the esophagogastroscopy and minimize the patients' dissatisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Patients with the indications for gastroduodenoscopy

Exclusion Criteria:

* Patients, who were receiving nonsteroidal anti-inflammatory drugs, pump inhibitors (PPI) or antibiotics in the last 3 weeks.
* Severe uncontrolled coagulopathy
* Prior history of gastric surgery.
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Procedure time | 4 months
  The time of examining the whole stomach was recorded, and the time for biopsy was not included.

SECONDARY OUTCOMES:
Patients' satisfaction | 4 months
  A 10-point scale was used to evaluate the patients' satisfaction (0 worst, 10 best). All the symptoms such as abdominal pain, distension and the like were all recorded.
  It is anticipated that the use of simethicone will significantly improve patients' satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, Principal Investigator — PLA General Hospital
Locations (1):
- PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Sajid MS, Rehman S, Chedgy F, Singh KK. Improving the mucosal visualization at gastroscopy: a systematic review and meta-analysis of randomized, controlled trials reporting the role of Simethicone +/- N-acetylcysteine. Transl Gastroenterol Hepatol. 2018 May 19;3:29. doi: 10.21037/tgh.2018.05.02. eCollection 2018. PMID 29971260
- [Derived] Sun X, Xu Y, Zhang X, Ma C, Li A, Yu H, Zhang W, Zhang H, Yang T, Miao X, Zhang H, Liu Y, Lu Z. Simethicone administration improves gastric cleanness for esophagogastroduodenoscopy: a randomized clinical trial. Trials. 2021 Aug 21;22(1):555. doi: 10.1186/s13063-021-05527-8. PMID 34419109